CLINICAL TRIAL: NCT06079749
Title: Risk of Chronic Post-surgical Pain After Simultaneous Versus Staged Bilateral Knee Arthroplasty: A Retrospective Study With Propensity Score Matching
Brief Title: Risk of Chronic Post-surgical Pain After TKA
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Do-Hyeong Kim, Professor, Gangnam Severance Hospital
Other Study IDs: 3-2023-0080
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Bilateral Total Knee Chronic Pain Following Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Simultaneous BTKA: Simultaneous BTKA
  Interventions: Procedure: Simultaneous BTKA
- Staged BTKA: Staged BTKA
  Interventions: Procedure: Staged BTKA

INTERVENTIONS:
Procedure: Simultaneous BTKA — Simultaneous BTKA
  Groups: Simultaneous BTKA
Procedure: Staged BTKA — Staged BTKA
  Groups: Staged BTKA

SUMMARY:
Chronic post-surgical pain (CPSP) is a common surgical complication. The role of timing in the development of CPSP after bilateral total knee arthroplasty (BTKA) is not well studied. We aimed to compare the occurrence of CPSP in patients who underwent simultaneous or staged BTKA without discharge between procedures.

ELIGIBILITY:
Inclusion Criteria:

* From October 12, 2012 to December 2, 2021, patients who underwent bilateral or staged knee replacement surgery during a single hospitalization under Professor Lee Woo-seok at the Department of Orthopedics at Gangnam Severance Hospital due to bilateral knee arthritis.

Exclusion Criteria:

* Patients whose post-operative pain information cannot be confirmed through outpatient visit records 1 year after surgery
* Those who have undergone surgery other than knee arthritis surgery within 1 year after surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From October 12, 2012 to December 2, 2021, patients who underwent bilateral or staged knee replacement surgery during a single hospitalization under Professor Lee Woo-seok at the Department of Orthopedics at Gangnam Severance Hospital due to bilateral knee arthritis.
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2012-10-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Chronic post-surgical pain at one year follow up | at one year follow up after surgery
  Numeric rating scale (0: no pain, 10: extreme pain)

IPD SHARING:
Plan to Share IPD: No